CLINICAL TRIAL: NCT00624182
Title: Phase 1 Study of Gemcitabine With Vaccine Therapy Targeting Tumor Antigen, URLC10, For The Patients With Unresectable or Recurrent Bile Duct Cancer
Brief Title: Gemcitabine With Peptide Vaccine Therapy in Treating Patients With Bile Duct Cancer
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Akita University Hospital (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Principal Investigator, Hiroshi Uchinami, Gastroenterological Surgery, Akita University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUGIS-001
Record Dates: First submitted 2008-02-19; First posted 2008-02-26 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Bile Duct Cancer
MeSH Terms: conditions — Bile Duct Neoplasms | interventions — Protein Subunit Vaccines; LY6K protein, human; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase I study (Experimental)
  Interventions: Biological: Peptide vaccine for URLC10; Drug: Gemcitabine

INTERVENTIONS:
Biological: Peptide vaccine for URLC10 — Increasing the doses of URLC10 peptides will be administered by subcutaneous injection on day 1, 8, 15, and 22 of each 28-day treatment cycles. Doses of 0.5, 1.0, 2.0mg/body are planned. Repeated cycles of this therapy will be continued until patients develop progressive disease or unacceptable toxicity, or maximum 2 cycles, whichever occurs first.
  Other Names: Gemcitabine
Drug: Gemcitabine — Gemcitabine will be administered intravenously at a fixed dose of 1000mg/m2 on day 1, 8, and 15. Repeated cycles of this therapy will be continued until patients develop progressive disease or unacceptable toxicity, or maximum 2 cycles, whichever occurs first.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and immune response of different doses of URLC10 peptide emulsified with Montanide ISA51 in combination with gemcitabine. Recommended phase II dose will be also determined.

DETAILED DESCRIPTION:
Our previous studies have demonstrated that up-regulated lung cancer 10 (URLC10) has been identified as a new target of tumor associated antigen using cDNA microarray technique combined with the expression profiles of normal and cancer tissues. We have also found that 100% of tissue samples from bile duct cancer express URLC10. We have determined the HLA-A*2402 and HLA-A*0201 restricted epitope peptides derived from URLC10.These epitope peptides have shown to induce specific Cytotoxic T Lymphocytes (CTL). Furthermore, 60% and 20% of Japanese population have HLA-A*2402 and HLA-A*0201, respectively. Therefore, these peptides are suitable for clinical trial. On the other hand, gemcitabine is a drug approved against bile duct cancer. Recent studies has reported that gemcitabine has an additional ability to improve immune response. From these results, synergistic effect between vaccine therapy and chemotherapy using gemcitabine will be expected.

In this clinical trial, we evaluate the safety, tolerability, and immune responses of different doses of URLC10 peptide emulsified with Montanide ISA51 as immunochemotherapy in the patients with unresectable or recurrent bile duct cancer. Toxicity profiles will be monitored, and antigen specific T cell responses will be described.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS

1. Advanced bile duct cancer precluding curative surgical resection and recurrent bile duct cancer
2. measurable disease by CT scan, ultrasonography, or other imaging modalities.

PATIENTS CHARACTERISTICS

1. ECOG performance status 0-2
2. Life expectancy >3 months
3. Laboratory values as follows 2,000/mm³< WBC < 15,000/mm³ Platelet count ≥ 75,000/mm³ Bilirubin ≤ 1.5 x the institutional normal upper limits AST, ALT, ALP ≤ 2.5 x the institutional normal upper limits Creatinine ≤ 1.5 x the institutional normal upper limits
4. HLA-A*2402 or HLA-A*0201
5. Able and willing to give valid written informed consent

Exclusion Criteria:

1. Pregnancy (women of childbearing potential: Refusal or inability to use effective means of contraception)
2. Breastfeeding
3. Serious or uncontrolled infection
4. Prior chemotherapy (except gemcitabine), radiation therapy, or immunotherapy within 4 weeks.
5. Other malignancy within 5 years prior to entry into the study
6. Concomitant treatment with steroids or immunosuppressing agent
7. Disease to the central nervous system
8. Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2008-02; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Safety (toxicities as assessed by NCI CTCAE version 3) | 5 years

SECONDARY OUTCOMES:
URLC10 peptide specific CTL induction | 5 years
DTH to URLC10 peptide | 5 years
Changes in levels of regulatory T cells | 5 years
Objective response rate as assessed by RECIST criteria | 5 years
Time to progression | 5 years
Survival rate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yuzo Yamamoto, MD, Study Chair — Department of Gastroenterological Surgery, Akita University, School of Medicine
Locations (1):
- Akita University Hosipital, Akita, Akita, Japan

REFERENCES:
- [Background] Date Y, Kimura A, Kato H, Sasazuki T. DNA typing of the HLA-A gene: population study and identification of four new alleles in Japanese. Tissue Antigens. 1996 Feb;47(2):93-101. doi: 10.1111/j.1399-0039.1996.tb02520.x. PMID 8851721
- [Background] Dauer M, Herten J, Bauer C, Renner F, Schad K, Schnurr M, Endres S, Eigler A. Chemosensitization of pancreatic carcinoma cells to enhance T cell-mediated cytotoxicity induced by tumor lysate-pulsed dendritic cells. J Immunother. 2005 Jul-Aug;28(4):332-42. doi: 10.1097/01.cji.0000164038.41104.f5. PMID 16000951
- [Background] Correale P, Cusi MG, Del Vecchio MT, Aquino A, Prete SP, Tsang KY, Micheli L, Nencini C, La Placa M, Montagnani F, Terrosi C, Caraglia M, Formica V, Giorgi G, Bonmassar E, Francini G. Dendritic cell-mediated cross-presentation of antigens derived from colon carcinoma cells exposed to a highly cytotoxic multidrug regimen with gemcitabine, oxaliplatin, 5-fluorouracil, and leucovorin, elicits a powerful human antigen-specific CTL response with antitumor activity in vitro. J Immunol. 2005 Jul 15;175(2):820-8. doi: 10.4049/jimmunol.175.2.820. PMID 16002679
- [Background] Suda T, Tsunoda T, Daigo Y, Nakamura Y, Tahara H. Identification of human leukocyte antigen-A24-restricted epitope peptides derived from gene products upregulated in lung and esophageal cancers as novel targets for immunotherapy. Cancer Sci. 2007 Nov;98(11):1803-8. doi: 10.1111/j.1349-7006.2007.00603.x. PMID 17784873
- [Background] Obama K, Ura K, Li M, Katagiri T, Tsunoda T, Nomura A, Satoh S, Nakamura Y, Furukawa Y. Genome-wide analysis of gene expression in human intrahepatic cholangiocarcinoma. Hepatology. 2005 Jun;41(6):1339-48. doi: 10.1002/hep.20718. PMID 15880566
- [Background] Marchand M, van Baren N, Weynants P, Brichard V, Dreno B, Tessier MH, Rankin E, Parmiani G, Arienti F, Humblet Y, Bourlond A, Vanwijck R, Lienard D, Beauduin M, Dietrich PY, Russo V, Kerger J, Masucci G, Jager E, De Greve J, Atzpodien J, Brasseur F, Coulie PG, van der Bruggen P, Boon T. Tumor regressions observed in patients with metastatic melanoma treated with an antigenic peptide encoded by gene MAGE-3 and presented by HLA-A1. Int J Cancer. 1999 Jan 18;80(2):219-30. doi: 10.1002/(sici)1097-0215(19990118)80:23.0.co;2-s. PMID 9935203
- [Background] Rosenberg SA, Yang JC, Schwartzentruber DJ, Hwu P, Marincola FM, Topalian SL, Restifo NP, Dudley ME, Schwarz SL, Spiess PJ, Wunderlich JR, Parkhurst MR, Kawakami Y, Seipp CA, Einhorn JH, White DE. Immunologic and therapeutic evaluation of a synthetic peptide vaccine for the treatment of patients with metastatic melanoma. Nat Med. 1998 Mar;4(3):321-7. doi: 10.1038/nm0398-321. PMID 9500606